CLINICAL TRIAL: NCT04152434
Title: Treatment of Chronic Migraine With Erenumab Alone or as an Add on Therapy; a Real World Prospective Observational Study
Brief Title: Treatment of Chronic Migraine With Erenumab Alone or as an Add on Therapy
Status: Completed | Type: Observational
Sponsor: Clinique des Céphalées de Montréal (Other)
Responsible Party: Principal Investigator, Guy Pierre Boudreau md, Medical Doctor, fellow in headache medecine, Clinique des Céphalées de Montréal
Other Study IDs: Erenumab 01
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Refractory Chronic Migraine
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Reduction in monthly migraine days all cohorts at 4 months: Migraineurs with 15-30 headache days per month at baseline were clustered in 3 categories. Failure of Erenumab was defined as no improvement in the frequency of monthly headache days. Group I: no preventive therapy, prior to the start of Erenumab. (No botox cohort). Group II: on Botulinum Toxin A (Botox), prior to the add on therapy with Erenumab. (Botox cohort).Group III: on an oral preventive drug, prior to the add on therapy with Erenumab. (No Botox cohort)
  Interventions: Drug: Erenumab Auto-Injector
- Selection of elegible paitients: A total of 158 patients were involved in this study. 118 patients (75%), received Erenumab 140 mg., and 40 patients (25%) received 70 mg. In the Botox cohort, of 650 patients, 90 (13%) patients were eligible. In the no Botox cohort, 533 patients, 83 (15%) patients were eligible.
  Interventions: Drug: Erenumab Auto-Injector
- Rate of adverse events related to Erenumab: 72 adverse events were experienced during the 4 months of treatment, mostly with the 140 mg. dose. The most frequent were: constipation 34%, fatigue 19%, itching 7.5%, muscle cramps 6.3%, increased headache 4.4%, rhinitis 4.4%, injection site discomfort 3.7%, lack of energy 3.1%
  Interventions: Drug: Erenumab Auto-Injector

INTERVENTIONS:
Drug: Erenumab Auto-Injector — Assess synergy of add on medication to Erenumab
  Other Names: Botox, and oral migraine preventives

SUMMARY:
Treatment of chronic migraineurs who have failed more than 3 preventive drugs with Erenumab alone, to reduce frequency of monthly migraine days or as an add on therapy

DETAILED DESCRIPTION:
The investigators treated chronic migraineurs that have failed more than 3 preventive drugs with Erenumab alone or as an add on therapy to: Reduce the frequency of monthly migraine days, to evaluate If the add on of Erenumab to another preventive therapy is superior to Erenumab alone, and assess all adverse events related to the use of Erenumab.

Migraineurs with 15-30 migraie days per month at baseline were clustered in 3 categories. Failure of Erenumab was defined as no improvement in the frequency of monthly migraine days. Group I: no preventive therapy, prior to the start of Erenumab. (No botox cohort). Group II: on Botulinum Toxin A (Botox), prior to the add on therapy with Erenumab. (Botox cohort).Group III: on an oral preventive drug, prior to the add on therapy with Erenumab. (No Botox cohort)

ELIGIBILITY:
Inclusion Criteria:

* chronic migraineurs with failure to more than 3 preventive treatments
* Naive to anti CGRP monclonal antibodies

Exclusion Criteria:

* episodic migraineurs,
* Other headache types

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with more than 15 migraine days per month, receiving Botox, or an oral preventive treatment, or without any preventive therapy. Have failed more than 3 preventive treatments previously
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in monthly migraine days | 5 months
  Change in frequency of monthly migraine days

SECONDARY OUTCOMES:
Change in frequency of monthly migraine days adding Erenumab to another preventive treatment, | 5 months
  Change in the frequency of monthly migraine days with Botox plus Erenumab,
Change in the frequency of monthly migraine days adding Erenumab to another preventive treatment | 5 months
  Change in the freqyency of monthly migraine days with an oral preventive plu erenumab
change in frequency of monthly migraine days with Erenumab alone | 5 months
  change in frequency of monthly migraine days without adding another preventive to Erenumab

CONTACTS AND LOCATIONS:
Overall Officials: Guy P Boudreau, md, Principal Investigator — Clinique des Céphalées de Montréal
Locations (1):
- Guy Pierre Boudreau, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No